CLINICAL TRIAL: NCT03087786
Title: Randomized, Parallel-Group, Assessor Blind Study To Evaluate Oral Mucosal Effects In Healthy Adult Smokers Associated With 3 Week Use Of Nicotine Bi-tartrate 4mg Mint Lozenges Relative To The Use Of Nicotine Polacrilex 4mg Mint Lozenges
Brief Title: Oral Mucosal Effects In Adult Smokers Associated With Two Nicotine Lozenge Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Niconovum USA (Industry)
Collaborators: Inflamax Research Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-NBTL-S-005
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Safety Issues
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotine Bitartrate 4mg Lozenge (Experimental): Nicotine Bitartrate Lozenge 4mg. Take 1 lozenge every 1-2 hours, as needed for 21 days
  Interventions: Drug: Nicotine Bitartrate Lozenge 4mg
- Nicotine Polacrilex 4mg Lozenge (Active Comparator): Nicotine Polacrilex Lozenge 4mg. Take 1 lozenge every 1-2 hours, as needed for 21 days
  Interventions: Drug: Nicotine Polacrilex 4Mg Lozenge

INTERVENTIONS:
Drug: Nicotine Bitartrate Lozenge 4mg — Test Product
  Other Names: Test Product
  Arms: Nicotine Bitartrate 4mg Lozenge
Drug: Nicotine Polacrilex 4Mg Lozenge — Active Comparator
  Other Names: Nicorette Lozenge 4mg
  Arms: Nicotine Polacrilex 4mg Lozenge

SUMMARY:
To study the oral mucosal effects in adult smokers associated with the use of two Nicotine Lozenge formulations.

DETAILED DESCRIPTION:
To assess the oral mucosal health associated with 3 weeks of use of test product, Nicotine Bitartrate 4 mg mint lozenge, relative to a reference product, Nicorette® [Nicotine Polacrilex] 4 mg mint lozenge, in healthy adult smokers motivated to quit smoking.

To evaluate the safety and tolerability of Nicotine Bitartrate 4 mg mint lozenge and Nicorette® [Nicotine Polacrilex] 4 mg mint lozenge in this subject population.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects who meet the following criteria at Screening may be included in the study.

1. Sex and Age: Males and females aged at least 18 years and older.
2. Informed of the nature of the study and have agreed to and are able to read, review, and sign the informed consent document prior to commencing any study specific procedures. The informed consent document will be written in English, therefore the volunteer must have the ability to read and communicate in English.
3. Must have smoked at least 10 cigarettes per day for the previous 12 months prior to screening.
4. Must smoke first cigarette within 30 minutes of waking up.
5. Must be motivated to quit smoking upon enrollment into the study.
6. Contraception: Females of childbearing potential who have been, in the opinion of the Investigator, practicing a reliable method of contraception for at least two months prior to study participation and must agree to remain on an acceptable method of contraception while participating in the study period using the study medication. Acceptable methods of contraception are hormonal birth control, intrauterine device, double barrier methods, vasectomized partner or abstinence.
7. Females of childbearing potential will be required to undergo a serum (Screening) and urine (Day 0) pregnancy test (must be negative).
8. Females of non-childbearing potential must be surgically sterile for at least three months prior to Screening or post-menopausal for at least two years.
9. General health: All study participants must have good general health and no impairment that would impede or affect ability to participate in the study as deemed acceptable by the Investigator.
10. Compliance: All study participants must understand and be willing to comply with all study procedures and restrictions.
11. Consent: All study participants must demonstrate willingness to participate as evidenced by voluntary written informed consent and must have received a signed and dated copy of the informed consent form.

Exclusion Criteria:

1. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
2. Nicotine use:

   1. Is unable/unwilling to stop using forms of tobacco (e.g., traditional cigarettes, chewing tobacco, nicotine gels, cigars, snuff tobacco, nicotine patch and electronic cigarettes) for the duration of the study.
   2. Is unable/unwilling to stop using other nicotine replacement therapy products throughout the duration of the study.
3. Disease: Has a medical history, which in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results, e.g., known history of heart disease, recent myocardial infarction or cerebrovascular accident (i.e., within 12 weeks prior to enrollment), unstable angina, severe cardiac arrhythmia, diabetes or peptic ulcer.
4. Demonstrates a reactive screen for Hepatitis B surface antigens, hepatitis C antibody, or HIV antibody.
5. Oral condition:

   1. Has history of oral surgery (including extractions) within four weeks of screening, operative dental work within seven days of screening, or a presence of any clinically significant oral pathology (as determined by an oral health professional - dentist or dental hygienist) including lesions, sores or inflammation of the mouth which would interfere with study assessments or confound the results.
   2. Has fixed retainers, orthodontic appliances, or either maxillary and/or mandibular dentures or other appliances which may interfere with the placement of the product.
   3. Has current or recurrent disease that could affect the site of application, the action, absorption of the study treatment, or clinical assessment.
   4. Has severe gingivitis, periodontitis or rampant caries (extensive dental decay, i.e., big/deep cavities, in many teeth), as diagnosed by an oral health professional- dentist or dental hygienist.
   5. Has the presence of oral or peri-oral ulceration including herpetic lesions at screening (subjects with these lesions may be re-examined at a subsequent appointment and may be able to be admitted at a later date if the ulceration or herpetic lesion heals) or Study Visit Day 0.
   6. Has elective dentistry scheduled during the study duration.
6. Allergy/Intolerance:

   1. Has a known or suspected intolerance or hypersensitivity to the study materials (or closely-related compounds) or any of their stated ingredients.
   2. Has a known genetic deficiency with an inability to metabolize aspartame or phenylalanine or has been diagnosed with phenylketonuria.
7. Clinical Study Participation:

   1. Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit at the start of the study.
   2. Previous participation in this study.
8. Substance abuse:

   1. Current or recent (within two years of screening) history of drug or alcohol abuse, misuse, physical or psychological dependence.
   2. Demonstrates a positive alcohol breath test.
   3. Demonstrates a positive urine drug screen without disclosure of corresponding prescribed concomitant medication(s) at Screening and Study Visit Day 0.
9. Urine glucose:

   a) Positive glucose urine screen.
10. Personnel:

    1. Is an employee of the Sponsor or the study site.
    2. Is a member of the same household as another subject in this trial.
11. Use of all over the counter (OTC) and prescription (Rx) lozenges after starting the study (Day 0 and onward).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-08-13 (Actual); Study Completion 2017-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, MD, CPI, Principal Investigator — Inflamax Research Incorporated
Locations (1):
- Inflamax Research Inc, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Started | 50 | 50
Completed | 48 | 50
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: One subject in the Nicotine Bitartrate group (Male, White, Age 21) was provided the study drug, but was then lost to followup. No evidence of ever taking any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (13.53) | 39.0 (10.94) | 39.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 29 | 31 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 41 | 43 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 39 | 69
  White | 19 | 11 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 50 | 99
Number of Particiapnts with OMI-20 Score of 0.00 [Number; unit: participants] — * Scale Title: The 20 Item Oral Mucositis Index (OMI-20)
  * The OMI-20 consists of nine items measuring erythema, nine measuring ulceration, one measuring atrophy, and one measuring edema; all are scored from 0 [none] to 3 [severe] and summed for a total possible score of 0-60.
  * A higher score means a worse outcome.
  * Only subjects without any oral pathology (as determined by an oral health professional - dentist or dental hygienist) including lesions, sores or inflammation of the mouth were included in the study (OMI-20 score of 0.00).
  participants | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: OMI-20 Total Score Change From Baseline to Day 3
Description: * Scale Title: The 20 Item Oral Mucositis Index (OMI-20)
  * The OMI-20 consists of nine items measuring erythema, nine measuring ulceration, one measuring atrophy, and one measuring edema; all are scored from 0 [none] to 3 [severe] and summed for a total possible score of 0-60.
  * A higher score means a worse outcome.
Time Frame: Day 3
Population: MITT: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 47 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.00)

2. Primary Outcome: OMI-20 Total Score Change From Baseline to Day 7
Description: as for outcome 1
Time Frame: Day 7
Population: MITT: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 49 | 50
score on a scale | 0.0 (0.00) | 0.0 (0.00)

3. Primary Outcome: OMI-20 Total Score Change From Baseline to Day 14
Description: as for outcome 1
Time Frame: Day 14
Population: MITT: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 48 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.00)

4. Primary Outcome: OMI-20 Total Score Change From Baseline to Day 21
Description: as for outcome 1
Time Frame: Day 21
Population: MITT: Modified Intent to Treat (no change in any participant was observed in the Nicotine Bitartrate arm)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 47 | 49
score on a scale | 0.00 (0.00) | 0.0 (0.20)

5. Secondary Outcome: OMI-20 Erythema Subscore Change From Baseline to Day 3
Description: * Scale Title: The 20 Item Oral Mucositis Index (OMI-20)
  * The OMI-20 contains a subset of nine items measuring erythema, all are scored from 0 [none] to 3 [severe], and summed for a total possible score of 0-27.
  * A higher score means a worse outcome.
Time Frame: Day 3
Population: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 47 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.00)

6. Secondary Outcome: OMI-20 Erythema Subscore Change From Baseline to Day 7
Description: as for outcome 5
Time Frame: Day 7
Population: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 49 | 50
score on a scale | 0.0 (0.00) | 0.0 (0.00)

7. Secondary Outcome: OMI-20 Erythema Subscore Change From Baseline to Day 14
Description: as for outcome 5
Time Frame: Day 14
Population: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 48 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.00)

8. Secondary Outcome: OMI-20 Erythema Subscore Change From Baseline to Day 21
Description: as for outcome 5
Time Frame: Day 21
Population: Modified Intent to Treat (no change in any participant was observed in the Nicotine Bitartrate arm)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 47 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.14)

9. Secondary Outcome: OMI-20 Ulcer Subscore Change From Baseline to Day 3
Description: * Scale Title: The 20 Item Oral Mucositis Index (OMI-20)
  * The OMI-20 contains a subset of nine items measuring ulcers, all are scored from 0 [none] to 3 [severe], and summed for a total possible score of 0-27.
  * A higher score means a worse outcome.
Time Frame: Day 3
Population: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 47 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.00)

10. Secondary Outcome: OMI-20 Ulcer Subscore Change From Baseline to Day 7
Description: as for outcome 9
Time Frame: Day 7
Population: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 49 | 50
score on a scale | 0.0 (0.00) | 0.0 (0.00)

11. Secondary Outcome: OMI-20 Ulcer Subscore Change From Baseline to Day 14
Description: as for outcome 9
Time Frame: Day 14
Population: Modified Intent to Treat (no change in any participant was observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 48 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.00)

12. Secondary Outcome: OMI-20 Ulcer Subscore Change From Baseline to Day 21
Description: as for outcome 9
Time Frame: Day 21
Population: Modified Intent to Treat (no change in any participant was observed in the Nicotine Bitartrate arm)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 47 | 49
score on a scale | 0.0 (0.00) | 0.0 (0.14)

13. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Count of the number of participants with Adverse Events.
Time Frame: Day 21
Population: Modified Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 49 | 50
Participants | 18 | 12

14. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Count of the number of participants with Serious Adverse Events
Time Frame: Day 21
Population: Modified Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

15. Secondary Outcome: Number of Participants Who Discontinued Due to Adverse Events (AEs)
Description: Count of the number of participants who discontinued due to Adverse Events.
Time Frame: Day 21
Population: Modified Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 days
Arm/Group | Nicotine Bitartrate 4mg Lozenge | Nicotine Polacrilex 4mg Lozenge
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 18/49 | 12/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Bitartrate 4mg Lozenge (N=49) | Nicotine Polacrilex 4mg Lozenge (N=50)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Dispepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Diarrhorea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Application Site Warmth (General disorders) | 0 (0) | 1 (1)
Vessel Puncture Site Bruise (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor and the PI have a Confidentiality Agreement stating:

* Each Party shall not disclose Confidential Information publicly or to any third party in an unauthorized manner.
* Each Party's obligations of confidentiality, non-disclosure and limited use imposed by this Agreement shall not apply to information or items that are required to be disclosed by governmental authority or by judicial process.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03087786/SAP_000.pdf
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03087786/Prot_001.pdf